CLINICAL TRIAL: NCT02994121
Title: Prospective Investigation of Multiple Sclerosis in the Three Rivers Region
Acronym: PROMOTE
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Zongqi Xia, MD, PhD, University of Pittsburgh
Other Study IDs: STUDY19080007
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, urine, saliva, and cerebrospinal fluid collection
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- People with Multiple Sclerosis or Related Disorders: Individuals must be 7 years or older, diagnosed with multiple sclerosis or related disorders, including a first central nervous system demyelinating episode with a positive MRI scan or abnormal MRI scans characteristic of MS but no clinical symptoms of the disease
- People without Multiple Sclerosis or Related Disorders: Control participants must be 7 years or older, have no known personal history of multiple sclerosis or related disorders, no other chronic disease, and can be a family member, unrelated household control, or control from the general population.

SUMMARY:
In this longitudinal prospective natural history study of multiple sclerosis (MS), the overarching goal is to understand the factors that influence individual variation in disease trajectory and treatment response and pave the way for realizing precision medicine in MS. Because MS is a chronic neurological disorder, this observational cohort study will span a 30-year time frame.

DETAILED DESCRIPTION:
Research Activities: Initial Questionnaire, Questionnaire for Self-Reported Outcomes, Biological Sample Collection (Blood, Stool, Urine, Cerebrospinal fluid), Genetic Analysis, Standard Quantitative Assessment of Function, Cognitive Assessment, Neuroimaging, Biometric Sensors, Social Network Questionnaire, Connor-Davidson Resilience Scale, NEO Five-Factor Inventory, and the COVID19 Response Surveys.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for MS patients include:

  1. Age 7 years or older
  2. Willing and able to provide consent (for >=18 years) or assent with permission from at least one of the child's parents (for <18 years)
  3. Diagnosis of multiple sclerosis or related disorders, including a first central nervous system demyelinating episode with a positive MRI scan or abnormal MRI scans characteristic of MS but no clinical symptoms of the disease
* For healthy controls:

  1. Age 7 years or older
  2. Willing and able to provide consent (for >=18 years) or assent with permission from at least one of the child's parents (for <18 years)
  3. No known personal history of multiple sclerosis or related disorders
  4. No other chronic diseases
  5. Family members, unrelated household controls, or controls from the general population could be eligible

There is no exclusion criteria.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People with multiple sclerosis and related disorders and controls
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2016-12; Primary Completion 2047-01 (Estimated); Study Completion 2047-01 (Estimated)

PRIMARY OUTCOMES:
Establish a prospective cohort of well-characterized MS patients and controls | within 30 years
  For this longitudinal prospective observational study, we will establish a prospective cohort of well-characterized MS patients and controls (2:1).
Investigate the predictors of the variations in disease trajectory and treatment response | within 30 years
  Understanding the factors that influence disease trajectory and treatment response will pave the way to realize precision medicine in delivering individualized MS care.

CONTACTS AND LOCATIONS:
Overall Officials: Zongqi Xia, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States